CLINICAL TRIAL: NCT01234844
Title: The Relationship Between Pet Therapy and "Well Being" in Geriatric Rehabilitation In-patients
Brief Title: The Relationship Between Pet Therapy and "Well-being" in Geriatric Rehabilitation In-patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MMC10157-2010CTIL; NCT01233466 (obsolete NCT alias)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Cerebrovascular Accident; Hip Fracture
Keywords: pet-therapy; guinea-pigs; rehabilitation; elderly
MeSH Terms: conditions — Stroke; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- care of guinea pigs (Other): Each patient serves as own control receiving "pet therapy "and "usual" occupational therapy on alternate days.
  Interventions: Behavioral: care of guinea pigs; Behavioral: guinea pigs

INTERVENTIONS:
Behavioral: care of guinea pigs — twice weekly sessions of care with guinea pigs
Behavioral: guinea pigs — twice weekly pet therapy and twice weekly "usual " occupational therapy

SUMMARY:
In -patients in a geriatric rehabilitation unit, will participate in structured therapy with guinea-pigs on the assumption that the therapy will reduce anxiety and improve the outcome of their rehabilitation.

DETAILED DESCRIPTION:
Measurement of anxiety before and after pet therapy using standardized questionaire.

ELIGIBILITY:
Inclusion Criteria:

willingness to touch the pets,-

Exclusion Criteria:

blindness,deafness,aphasia, lack of knowledge of hebrew language,allergy or phobia to animals.MMSE less than 21,duration of admission lessthan two weeks.-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The relationship between pet-therapy and "well-being"among geriatric rehabilitation in-patients | two weeks
  use of validated questionaires to measure mood,anxiety and quality of life before and after the pet therapy

SECONDARY OUTCOMES:
anxiety score | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Devorah T Spiegel, MB.ChB, Principal Investigator — Meir Hospital
Locations (1):
- Geriatric Department ,Meir Hospital, Kfar Saba, Israel